CLINICAL TRIAL: NCT02097654
Title: A Prospective, Multinational, Randomized, Open Label Parallel Arm Trial With Blinded Outcome Adjudication Quantifying the Efficacy of SENATOR in Reducing Adverse Drug Reactions in Older Hospitalized Subjects
Brief Title: Clinical Trial of a New Software ENgine for the Assessment & Optimization of Drug and Non-drug Therapy in Older peRsons
Acronym: SENATOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Clanwilliam Health (Unknown); University of East Anglia (Other); ARTTIC International Management Services (Unknown); Clininfo S.A. (Industry); NHS Grampian (Other Government); University Ghent (Other); Hospital Universitario Ramon y Cajal (Other); Istituto Nazionale di Ricovero e Cura per Anziani (Other); Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Denis O'Mahony, Professor, Department of Medicine, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRF-C-12-05
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Adverse Drug Reactions
Keywords: Hospital acquired; Elderly
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Block randomized parallel arm trial.
Who Masked: Outcomes Assessor
Masking Description: For outcome data, details were extracted from patients' case records to determine if trigger list adverse clinical events had occurred following randomization. These trigger list events represented the great majority of adverse drug reactions (ADRs) and were independently adjudicated by a blinded end-point committee comprised of the co-PI's, such that no co-PI adjudicated potential ADRs at his own site.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SENATOR (Experimental): Physicians attending multi-morbid older patients i.e. with 3 or more chronic medical conditions receive a SENATOR software-generated report with advice details on potentially inappropriate pharmacotherapy and/or potentially inappropriate prescribing omissions.
  Interventions: Other: SENATOR software generated pharmacotherapy advice report.
- Control (No Intervention): Standard pharmaceutical care as per local practice.

INTERVENTIONS:
Other: SENATOR software generated pharmacotherapy advice report.
  Arms: SENATOR

SUMMARY:
Primary Objective: To quantify the benefits of the SENATOR decision support software on the reduction of ADR rates in older hospitalized patients. Secondary Objectives: To evaluate the effect of SENATOR with regard to use of appropriate non-pharmacological therapies in subjects with one core geriatric syndrome.

Tertiary Objectives: to examine the association of SENATOR use with subject survival, morbidity and health related quality of life.

Health Economic Objective: To examine the potential health economic consequences of using SENATOR.

There are two study phases:

Phase I: Prospective multinational, multicentre observational study to estimate the baseline adjudicated medical and surgical ADR rates by clinical subspeciality in 6 international sites.

Phase II: Prospective multinational, multicentre, block randomized, two parallel arm, open label, controlled trial, with blinded outcome ascertainment, of the efficacy of SENATOR software in reducing ADRs in older hospitalized subjects.

DETAILED DESCRIPTION:
Phase I is designed to test the electronic case report form (eCRF) and the ADR ascertainment method in the six clinical sites in advance of Phase II (randomization phase).

In Phase I, we recruited 644 older multi-morbid patients from the 6 clinical sites. After obtaining written informed consent, patients' demographic, clinical and medication details were entered to the eCRF. In the event of one a 12 item Trigger List of adverse clinical events occurring, the eCRF automatically generated a Trigger List assessment proforma. The 12 items in the Trigger List included:

1. New onset falls
2. New onset unsteady gait
3. Acute kidney injury
4. Symptomatic orthostatic hypotension
5. Serum electrolyte disturbance
6. Symptomatic bradycardia
7. New onset major constipation
8. Acute bleeding
9. Acute dyspepsia/nausea/vomiting
10. Acute diarrhea
11. Delirium
12. Symptomatic hypoglycemia

In addition, we have included 'Unspecified adverse event' in order to capture the wide range of well recognized ADRs associated with various medications. For example, the rapid onset of a generalized maculopapular rash in a patient with penicillin hypersensitivity would be identified as an ADR under the 'Unspecified adverse event' category.

ADR adjudication in Phase I was blinded and no ADR adjudications were undertaken by the site principal investigator (PI). ADRs were defined as 'definite', probable', 'possible', 'unlikely' or 'indeterminate' according to WHO-UMC ADR causality critria. ADR severity was defined according to a modified Hartwig ADR severity scale ranging from Level 1 (trivial) to Level 7 (fatal).

Consensus on ADR causality was achieved through a potential endpoint adjudication committee (PEPAC), whose members were the 6 clinical site PI's. A matrix for achieving consensus was devised, such that there was a final decision on the causality of all potential ADRs.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent by the patient or legal guardian/next-of-kin
2. Age ≥ 65 years
3. Arrival to hospital within previous 72 hours
4. Admitted as a general medical or surgical on call patient
5. Anticipated in-hospital stay of > 48 hours,
6. ≥ 3 active (requiring current medication) chronic medical disorders

Exclusion Criteria:

1. Admitted under:

   * Geriatric Medicine
   * Clinical Pharmacology
   * Palliative Medicine
   * Clinical Oncology
   * Hematology
2. Intention of primary team at the time of subject admission to seek a Geriatric Medicine, Clinical Pharmacology or Palliative Medicine in-patient consultation
3. Life expectancy in the opinion of the admitting clinician of < 3 months
4. Admission directly to an intensive care unit,
5. Admission with primary acute psychiatric illness (excluding delirium)
6. Admission with non-accidental overdose/self-harm
7. Anticipated immediate transfer to alternative non-participating clinical service/hospital
8. Clinical diagnosis of acute Liver failure
9. estimated Glomerular Filtration Rate <10 ml/min per 1.73 m2
10. Solid organ transplant recipients
11. Patients with malignancy receiving systemic chemotherapy
12. Hospitalized for elective procedure
13. Patient was more than 24 hours in the Emergency Department under the care of a different team to that which finally is in charge of them
14. Patients who are actively participating in another clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Incident adverse drug reactions (ADRs). at least one likely or certain, non-trivial hospital acquired ADR. | Day 14 of hospital stay or discharge, which ever comes first
  Subjects adjudicated by the Potential Endpoint Committee as having experienced one or more probable or certain adverse drug reactions (ADRs).

CONTACTS AND LOCATIONS:
Overall Officials: Joesph Eustace, MD FRCPI, Study Director — University College Cork, Ireland; Antonio Cherubini, MD PhD, Principal Investigator — IRCCS-INRCA Ancona, Italy; Adalsteinn Gudmundsson, MD PhD, Principal Investigator — Landspitali University Hospital, Iceland; Alfonso Cruz-Jentoft, MD, Principal Investigator — Hospital Universitario Ramōn y Cajal Madrid; Roy Soiza, MD FRCP, Principal Investigator — NHS Grampian, Aberdeen, Scotland; Mirko Petrovic, MD PhD, Principal Investigator — Ghent University Hospital, Ghent, Belgium; Denis O'Mahony, MD FRCPI, Study Chair — University College Cork, Ireland
Locations (1):
- University College Cork, Cork, Munster, Ireland

REFERENCES:
- [Derived] Dalton K, Curtin D, O'Mahony D, Byrne S. Computer-generated STOPP/START recommendations for hospitalised older adults: evaluation of the relationship between clinical relevance and rate of implementation in the SENATOR trial. Age Ageing. 2020 Jul 1;49(4):615-621. doi: 10.1093/ageing/afaa062. PMID 32484853
- [Derived] Lavan AH, O'Mahony D, Gallagher P, Fordham R, Flanagan E, Dahly D, Byrne S, Petrovic M, Gudmundsson A, Samuelsson O, Cherubini A, J Cruz-Jentoft A, Soiza RL, Eustace JA. The effect of SENATOR (Software ENgine for the Assessment and optimisation of drug and non-drug Therapy in Older peRsons) on incident adverse drug reactions (ADRs) in an older hospital cohort - Trial Protocol. BMC Geriatr. 2019 Feb 13;19(1):40. doi: 10.1186/s12877-019-1047-9. PMID 30760204
- See also: Development and clinical trial of a new Software ENgine for the Assessment & Optimization of drug and non-drug Therapy in Older peRsons (SENATOR). — http://www.senator-project.eu